CLINICAL TRIAL: NCT00758992
Title: Peripheral Blood Stem Cells Obtained From Normal Volunteers for Studying Retroviral Vector Mediated Gene Transfer Into Primitive Hematopoietic Cells and Vector Mediated Transgene Expression in Mature Hematopoietic Lineages
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PBSCRV; P01HL053749 (NIH); 2010037 (Other: Doris Duke Foundation)
Record Dates: First submitted 2008-09-18; First posted 2008-09-25 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Immunodeficiency
Keywords: gene transfer
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Immunodeficient mice: Please see the Study Description for complete information.

SUMMARY:
These studies are designed to evaluate the relative efficiency of gene transfer into primitive human hematopoietic cells by comparing lentiviral and foamy virus vectors as vehicles for transfer and expression of globin genes. Normal volunteers will serve as research participants. Each will receive a 4 day course of Granulocyte-Colony Stimulating Factor (G-CSF) after which a peripheral blood apheresis will be performed to recover a mononuclear cell population enriched in primitive hematopoietic cells. The stem and progenitor cells will be purified by selection based on expression of the CD34 antigen. The CD34+ population will be cultured in vitro with various cytokines and transduced with vector particles. The efficiency of gene transfer will be evaluated in the transduced CD34+ population, in progenitors contained within that population by culture in semisolid media and in cells capable of establishing human hematopoiesis in immunodeficient mice. The level of transgene expression will be evaluated in mature hematopoietic lineages that develop in vitro or in immunodeficient mice.

DETAILED DESCRIPTION:
The peripheral blood has been established as a source of hematopoietic stem cells, providing an alternative source to bone marrow for hematopoietic reconstitution of patients with oncologic, hematologic, and genetic diseases. Although apheresis is less efficient than bone marrow harvesting for collection of large numbers of CD34+ (a marker of early hematopoietic precursors) cells, apheresis is less traumatic, requires no anesthesia and can be performed more frequently than bone marrow harvesting. The purpose of this preclinical research project is to investigate the use of hematopoietic stem cells mobilized into peripheral blood as targets for retroviral-mediated gene therapy, to compare the efficiency of transduction of primitive cells with the lentiviral and foamy viral vector systems and to evaluate the ability to expand those stem cells ex vivo using hematopoietic growth factors (cytokines). Research participants in this study will be healthy adult volunteers.

The growth factor, Granulocyte-Colony Stimulating Factor (G-CSF), will be given for 4 days prior to apheresis to mobilize increased numbers of primitive hematopoietic cells from the bone marrow into the circulation. Nucleated blood cells will be collected by apheresis and a CD34+-enriched cell population isolated using antibody-based techniques.

Administration of G-CSF is essential to allow collection of sufficient numbers of primitive stem and progenitor cells from normal volunteers. In the dose to be used in this study, a 15-35 fold increase in the concentration of CD34+ cells occurs in peripheral blood over the 4 days of G-CSF administration resulting in an apheresis product which contains, on average, about 1-2 x1010 nucleated cells from which 1-2x108 purified CD34+cells can be recovered. This number is sufficient to allow an experimental design which includes in vitro culture, transduction with vector particles and assay of transduced cells in the immunodeficient mouse model.

The use of G-CSF for mobilization of stem and progenitor cells is a widely used clinical technique for both autologous and allogeneic transplantation which has proved both safe and effective. Bone and muscle pain, headache and fatigue are the most common complications which are typically managed with acetaminophen and rarely require discontinuation of G-CSF. Transient elevations in alkaline phosphatase and LDH are common. Follow-up studies have shown prolonged, mild neutropenia, lymphopenia and thrombocytopenia following G-CSF administration and apheresis. Splenic enlargement has been shown by non-invasive measurements and four cases of splenic rupture in normal individuals have been described. A reduction in arterial pO2 associated with a decrease in the O2 saturation from 98 to 96% has been reported. Transient thrombophilia has been inferred based on changes in blood coagulation parameters.

Other rare complications have been reported including the development of inflammatory or infectious lesions. A fatal crisis occurred in a sibling donor for allogeneic transplantation who had hemoglobin SC disease. These rare complications should be put in the context that G-CSF administration followed by apheresis to recover primitive hematopoietic cells from normal individuals has been utilized in all major transplant centers for more than a decade and has generally been safe and without significant complications. We propose to minimize the risk of serious complications by limiting the age range of research participants to 18-40 years and excluding those with a history of inflammatory disease, cardiovascular disease, thrombosis or pulmonary embolization, inflammatory skin disorders, hematological disease or hemoglobinopathy.

The ability to expand mobilized CD34+ cells in vitro using various cytokine combinations and culture conditions will be examined using flow cytometry, in vitro colony assays and by quantitating the concentration of cells that are able to establish hematopoiesis in immunodeficient mice. Both unexpanded and expanded CD34+ cells will be used in experiments designed to investigate their suitability as targets for retroviral-mediated gene transfer. Gene transfer efficiency and functional expression of transferred sequences will be assessed in the differentiated progeny of CD34+ cells.

We plan to compare the lentiviral and foamy virus vector systems with respect to relative efficiency of gene transfer into primitive human hematopoietic cells. Various substances e.g., Fibroblast Growth Factor -1 and Wnt 3A, that have been reported to cause expansion of primitive murine hematopoietic cells will also be evaluated for their effects of primitive human hematopoietic cells in culture. Another focus is the comparison of various globin gene vectors with respect to the relative levels of globin gene expression in differentiating erythroid cells. Finally, the impact of cryopreservation on viability and engraftment potential of primitive hematopoietic cells will be assessed. This research proposal will provide preclinical data that will aid in the development of treatment strategies for genetic diseases, specifically hemoglobin disorders, based on gene transfer into repopulating stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years and less than or equal to 40.
* Meets donation criteria for autologous blood donors per SJCRH Blood Donor Center standard operating procedure.
* Adequate venous access for apheresis on examination as per the judgment of the Blood Donor Center nursing staff, physician staff or physician investigators.

Exclusion Criteria:

* Females - lactating.
* Concurrent use of systemic medications that in the judgment of the physician investigators adversely affect platelet function, such as aspirin or non-steroidal antiinflammatory agents.
* Any of the following diagnoses (prior or current):

  * pulmonary disease.
  * inflammatory disorder.
  * coronary artery disease.
  * stroke (cerebral vascular accident).
  * hypertension.
  * cardiac arrhythmias.
  * venous thrombosis.
  * pulmonary embolus
  * hematological disease.
  * eczema or psoriasis.

Additional eligibility criteria (to be obtained after signing informed consent)

* Body mass index less than 30 kg/m2.
* No hepatomegaly or splenomegaly.
* Hemoglobin greater than or equal to 12.5 g/dL.
* Platelet count greater than or equal to 150,000/mm3.
* Total WBC > 4200/ul and neutrophil count >1800/ul.
* Females - not pregnant (negative serum or urine; to be obtained after signing informed consent).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Adult Research Participants
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To compare the relative efficiencies of lentiviral and foamy virus vectors in transducing primitive hematopoietic cells mobilized into peripheral blood by cytokine administration. | Up to 3 years after apheresis collection of donor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur W Nienhuis, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols